CLINICAL TRIAL: NCT06902974
Title: A Phase 2, Open-Label Study Investigating the Safety and Efficacy of Psilocybin-Assisted Therapy for Sexual Assault-Related Posttraumatic Stress Disorder (PTSD)
Brief Title: Psilocybin-Assisted Therapy for Sexual Assault-Related PTSD
Acronym: SUN004
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunstone Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2025-02-25; First posted 2025-03-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-03

CONDITIONS: Post Traumatic Stress Disorder; PTSD
Keywords: PTSD; sexual assault; psilocybin; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, single-center, fixed dose, open-label study to explore the efficacy, safety, and tolerability of a 25 mg dose of oral psilocybin with therapy in adult cisgender women participants with PTSD secondary to an index trauma of sexual assault.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin-Assisted Therapy (Experimental): This is a Phase 2, single-center, fixed dose, open-label study to explore the efficacy, safety, and tolerability of a 25 mg dose of oral psilocybin with therapy in adult cisgender women participants with PTSD secondary to an index trauma of sexual assault. There is no comparator group.
  Interventions: Drug: Psilocybin 25 mg

INTERVENTIONS:
Drug: Psilocybin 25 mg — Single dose, 25mg psilocybin, encapsulated, oral administration
  Other Names: Psilocybin-assisted therapy

SUMMARY:
The proposed Phase 2, single-center, fixed dose, open-label study will explore the efficacy, safety, and tolerability of 25 mg dose of oral psilocybin in conjunction with therapy in cisgender women participants diagnosed with PTSD secondary to an index trauma of sexual assault.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women who are at least 18 years old.
* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for current PTSD secondary to sexual assault (i.e., index trauma is sexual assault that occurred 6 or more months in the past).
* CAPS-5 score of 25 or higher at Baseline.
* Are able to swallow pills.
* Are willing to be driven home after the Dosing Session with a family member or caregiver or trusted transportation.
* Are able to complete all protocol-required assessment tools without any assistance or alteration to the copyrighted assessments, and to comply with all study visits.
* If able to become pregnant (i.e., with uterus and associated reproductive organs, fertile, following menarche and until becoming post-menopausal unless permanently sterile), must have a highly sensitive negative pregnancy test at study entry and prior to the Dosing Session, and must agree to use adequate birth control through 10 days after the Dosing Session if sexually active with a biologically male partner. Adequate birth control methods include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e. condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom).
* Must agree to inform the clinical investigators within 48 hours of any medical conditions and procedures.
* Are proficient in speaking and reading English.
* Agree to have all clinic visit sessions recorded to audio and/or video. Participants may opt out of the data analysis of the recordings.
* Agree to the following lifestyle modifications: a light breakfast 2 to 3 hours before dosing is permitted, however, participants will refrain from caffeine and nicotine 2 hours prior to dosing sessions and at least 6 hours after dosing, abstain from alcohol for 24 hours prior to dosing, not enroll in any other interventional clinical studies during the duration of the study, be driven home after the Dosing Session, and commit to medication dosing, therapy, and study procedures.
* Agree to refrain from beginning new medication and/or psychotherapy treatment.
* Continued treatment with SSRIs will be permitted if participants have been on a stable dose for 3 months or longer prior to enrollment. However, participants must be tapered off of monoamine oxidase inhibitors (MAOIs) prior to dosing.

In addition, participants may remain in stable (> 3 months) psychotherapy.

* May have well-controlled hypertension that has been successfully treated with anti-hypertensive medicines.
* May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
* May have alcohol or substance use disorder if participant is not in withdrawal or requiring detox. Participants must have a plan, agreed upon by the principal investigator or designated physician, to reduce use of alcohol or other substances and to manage symptoms without self-medicating. Enrollment will require that, in the judgment of the principal investigator or designated physician, the plan for decreasing substance use is realistic and has a good chance of succeeding in order to prevent substance use from impacting the safety or efficacy of the investigational treatment.
* May have a history of or current Diabetes Mellitus (Type 2) if additional screening measures rule out underlying cardiovascular disease, if the condition is judged to be stable on effective management, and with approval by the principal investigator or designated physician.
* May have hypothyroidism if taking adequate and stable thyroid replacement medication.

Exclusion Criteria:

* Male
* Condition impairing oral intake or digestive absorption.
* Are not able to give adequate informed consent.
* Significant suicide risk as defined by suicidal ideation with intend and a plan as endorsed on items 5 on the C-SSRS within the past 3 months
* Have any current problem which, in the opinion of the principal investigator or designated physician, might interfere with participation.
* Would present a serious risk to others as established through clinical interview and contact with treating therapist.
* Have a history of, or a current primary, schizophrenia, schizoaffective disorder or any form of psychotic disorder, major depressive disorder with psychotic features, bipolar affective disorder type 1, or personality disorders.
* Require ongoing concomitant therapy with a psychiatric medication with exceptions described below (see Section 6.6).
* Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment.
* Have evidence or history of recent stroke (< 6 months from signing of ICF), recent myocardial infarction (< 6 months from signing of ICF), or clinically significant arrhythmia within 1 year of signing the ICF.
* Have evidence or history of significant (controlled or uncontrolled) hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder, or any other medical disorder judged by the investigator to significantly increase the risk of psilocybin administration.
* Have uncontrolled hypertension using the standard criteria of the American Heart Association (values of 140/90 milligrams of Mercury [mmHg] or higher).
* Abnormal and clinically significant results on vital signs, ECG, or laboratory tests at screening and baseline
* Have symptomatic liver disease.
* Are pregnant, nursing, or able to become pregnant and are not practicing an effective means of birth control if sexually active with a biologically male partner.
* Have hypersensitivity to any ingredient of the study drug.
* Positive urine drug screen for illicit drugs or drugs of abuse prior to the Dosing Session. Any positive urine drug test will be reviewed with participants to determine the pattern of use and eligibility will be determined at the investigator's discretion.
* Current enrollment in any investigational drug or device study or participation in such within 30 days of screening.
* Other personal circumstances and behavior judged to be incompatible with establishment of rapport or safe exposure to psilocybin or completion of clinical study procedures (e.g., active participation in legal proceedings).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender femal
Enrollment: 35 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of psilocybin-assisted therapy in adult participants with PTSD secondary to sexual assault | Between ICF until End of Study (approx. 8 weeks from baseline)
  Incidence and occurrence of treatment emergent adverse events (TEAEs) and SAEs from signing of Informed Consent Form (ICF) until the End of Study (EOS) Visit
To assess the safety and tolerability of psilocybin-assisted therapy in adult participants with PTSD secondary to sexual assault | Between Baseline to End of Study (approx. 8 weeks from baseline)
  Incidence of changes in suicidal ideation/behavior (measured using the C-SSRS) score at all visits from Baseline to End of Study Visit

SECONDARY OUTCOMES:
To assess the efficacy of psilocybin-assisted therapy on symptoms of PTSD in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from baseline)
  Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total score
  The CAPS is the gold standard in PTSD assessment. The CAPS-5 is a 30-item structured interview that can be used to:
  Make current (past month) diagnosis of PTSD Make lifetime diagnosis of PTSD Assess PTSD symptoms over the past week In addition to assessing the 20 DSM-5 PTSD symptoms, questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization).
  Scores can range from 0 (absent) - the respondent denied the problem or the respondent's report doesn't fit the DSM-5 symptom criterion" to 4 (extreme/incapacitating) "The respondent described a dramatic symptom, far above threshold.'
To assess the efficacy of psilocybin-assisted therapy on symptoms of PTSD in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from baseline)
  Change in the PTSD Checklist (PCL-5)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD.
  Interpretation of the PCL-5 should be made by a clinician. The PCL-5 can be scored in different ways:
  A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items.
  DSM-5 symptom cluster severity scores can be obtained by summing the scores for the items within a given cluster, i.e., cluster B (items 1-5), cluster C (items 6-7), cluster D (items 8-14), and cluster E (items 15-20).
  A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 B item (questions 1-5), 1 C item (questions 6-7), 2 D items (questions 8-14), 2 E items (questions 15-20).
To assess the efficacy of psilocybin-assisted therapy on symptoms of PTSD in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from baseline)
  Change in State-Trait Anxiety Inventory (STAI) The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress (e.g., Greene et al., 2017, Ugalde et al., 2014).
  Form Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
To assess the efficacy of psilocybin-assisted therapy on symptoms of PTSD in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from baseline)
  Change in Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR-16) total score
  The Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR16) is a 16-item self-report questionnaire used to assess the severity of depressive symptoms, with scores ranging from 0 to 27, indicating no to very severe depression.
To assess the efficacy of psilocybin-assisted therapy on symptoms of PTSD in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from baseline)
  Time to event measures: starting of antidepressant medication for any reason, starting medication for continuing PTSD or depressive symptoms, relapse from a previously recovered state (clinician judgement, supported by the PCL-5), and onset or worsening of any psychiatric symptoms. Participants who withdraw from the study will be censored from the time to event analysis.
To assess the effect of psilocybin-assisted therapy on quality of life and participant functional impairment in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from Baseline)
  Change from Baseline to EOS in the Sheehan Disability Scale (SDS) total score.
  The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
  How to Score Total score 0-30 (0 unimpaired, 30 highly impaired) Work/school (0-10) Social life (0-10) Family life/home responsibilities (0-10 Scores of ≥5 on any of the 3 scales; high scores are associated with significant functional impairment.
To assess the effect of psilocybin-assisted therapy on quality of life and participant functional impairment in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from Baseline)
  Change from Baseline to EOS in the EuroQoL-5 Dimension, 5 level Scale (EQ-5D-5L) total score
  The EuroQoL 5-Dimension, 5-level Scale (EQ-5D-5L) is a health-related quality of life (HRQoL) questionnaire that assesses health status across five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) using a 5-level scale for each dimension, ranging from no problems to extreme problems.
To assess the effect of psilocybin-assisted therapy on quality of life and participant functional impairment in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from Baseline)
  Proportion of participants with clinical response in CAPS-5 total score from Baseline. Clinical response in CAPS-5 is defined in a reduction of 10 or more points.
To assess the effect of psilocybin-assisted therapy on quality of life and participant functional impairment in adult participants with PTSD secondary to sexual assault | From Baseline to End of Study (approx. 8 weeks from Baseline)
  Proportion of participants achieving remission of PTSD symptoms as measured by the CAPS-5 following the Dosing Session. Clinical remission is defined as a Loss of Diagnosis plus a severity score < 20.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Agrawal, MD, MSC, Principal Investigator — Sunstone Medical, PC
Locations (1):
- Sunstone Medical, PC, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing not required